CLINICAL TRIAL: NCT00926809
Title: Helicobacter Pylori Eradication Therapy on the Healing of Iatrogenic Gastric Ulcer After Endoscopic Mucosal Resection of Gastric Neoplastic Lesions: a Multicenter, Randomized, Double Blind, and Placebo Controlled Trial
Brief Title: H. Pylori Eradication on Healing of Iatrogenic Gastric Ulcer by Endoscopic Mucosal Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean College of Helicobacter and Upper Gastrointestinal Research (Other)
Responsible Party: Ho June Song, Korean College of Helicobacter and Upper Gastrointestinal Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009KHR001
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Ulcer
Keywords: endoscopic mucosal resection; iatrogenic
MeSH Terms: conditions — Ulcer | interventions — Lansoprazole; Proton Pump Inhibitors; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eradication (Active Comparator): Helicobacter pylori eradication
  Interventions: Drug: Lansoprazole (proton pump inhibitor), amoxicillin, clarythromycin
- No eradication (Placebo Comparator): No eradication for Helicobacter pylori
  Interventions: Drug: Lansoprazole (proton pump inhibitor), placebo

INTERVENTIONS:
Drug: Lansoprazole (proton pump inhibitor), amoxicillin, clarythromycin — Lansoprazole, Amoxicillin 1000 mg, Clarithromycin 500 mg
  Arms: Eradication
Drug: Lansoprazole (proton pump inhibitor), placebo — Lansoprazole, Amoxicillin placebo, Clarythromycin placebo
  Arms: No eradication

SUMMARY:
This study will evaluate the effect of Helicobacter pylori eradication therapy on the healing of iatrogenic gastric ulcer caused by endoscopic mucosal resection of gastric neoplastic lesions and is a multicenter, randomized, double blind, and placebo controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* 30 - 75 years old
* Early gastric cancer (< 3 cm in size, mucosa confined, differentiated type) or gastric adenoma (< 3 cm in size)
* Helicobacter pylori positive

Exclusion Criteria:

* Medication of anti-secretory drugs (proton pump inhibitors, H2-receptor antagonists, antacid, bismuth compound)
* History of Helicobacter pylori eradication
* History of gastric surgery or other cancers
* Major comorbidities
* Medication of ASA, NSAIDS, steroids, anti-coagulants

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
ulcer healing rate by endoscopic assessment | 8 weeks

SECONDARY OUTCOMES:
ulcer reduction rate by endoscopic assessment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Chae Jung, Principal Investigator — Korean College of Helicobacter and Upper Gastrointestinal Research
Locations (6):
- South Korea (6):
  - National Cancer Center Korea, Goyang
  - Asan Medical Center, Seoul
  - Korea University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul